CLINICAL TRIAL: NCT01994733
Title: Two phosphAte taRGets in End-stage Renal Disease Trial (TARGET): Intensive vs Liberalized Phosphate Control in Hemodialysis Recipients
Brief Title: Two phosphAte taRGets in End-stage Renal Disease Trial (TARGET)
Acronym: TARGET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ron Wald, Staff Physician, Division of Nephrology; Scientist, Li Ka Shing Knowledge Institute of St. Michael's Hospital, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: End-stage Renal Disease
Keywords: end-stage renal disease; hemodialysis; mineral metabolism; serum phosphate; phosphate binders
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive phosphate control (Experimental): Individuals randomized to this arm will be exposed to a treatment strategy that targets a P of < 1.50 mmol/L, reflecting the recommendations of current guidelines. Titration of the calcium carbonate dose will be the core of this approach and this will be complemented by usual recommendations regarding dietary P restriction. Dietitians will be available to provide counseling with regards to any aspect of the end-stage renal disease diet, as per usual dialysis unit practice.
  Interventions: Drug: Calcium carbonate ( Intensive phosphate control)
- Liberalized phosphate control (Active Comparator): Individuals in this arm will be exposed to a treatment strategy that allows P to rise above 2.00 mmol/L. This will be accomplished through structured reduction of P binders already in use (as per the algorithm detailed below). "Rescue" P binding will be instituted if P rises above 2.50 mmol/L. Dietitians will be available to provide counseling regarding any aspect of the end-stage renal disease diet, as per usual dialysis unit practice, but will not provide counseling on dietary P restriction unless the P rises above 2.50 mmol/L.
  Interventions: Drug: Calcium carbonate (Liberalized phosphate control)

INTERVENTIONS:
Drug: Calcium carbonate ( Intensive phosphate control) — Individuals randomized to this arm will be exposed to a treatment strategy that targets a P of < 1.50 mmol/L, reflecting the recommendations of current guidelines. Titration of the calcium carbonate dose will be the core of this approach and this will be complemented by usual recommendations regarding dietary P restriction. Dietitians will be available to provide counseling with regards to any aspect of the end-stage renal disease diet, as per usual dialysis unit practice
  Other Names: Calcium carbonate
  Arms: Intensive phosphate control
Drug: Calcium carbonate (Liberalized phosphate control) — Individuals in this arm will be exposed to a treatment strategy that allows P to rise above 2.00 mmol/L. This will be accomplished through structured reduction of P binders already in use (as per the algorithm detailed below). "Rescue" P binding will be instituted if P rises above 2.50 mmol/L. Dietitians will be available to provide counseling regarding any aspect of the end-stage renal disease diet, as per usual dialysis unit practice, but will not provide counseling on dietary P restriction unless the P rises above 2.50 mmol/L.
  Arms: Liberalized phosphate control

SUMMARY:
Patients with end-stage renal disease (ESRD) who have elevated serum phosphate (P) levels have significantly higher mortality rates compared to those with normal P. In patients receiving conventional dialysis regimens, serum P may be lowered through dietary intervention and use of P binders, though these have potentially important side effects and may adversely impact quality of life. Whether lowering P, and / or targeting specific P levels improve survival and clinical outcomes is unknown. Despite this uncertainty, over 90% of patients with ESRD receive P lowering therapy and guidelines for the care of patients with ESRD are increasingly calling for more aggressive phosphate lowering. This intensive P lowering results in extra medications (and their associated side-effects), and higher health care costs. We are uncertain whether the intensification of P control results in measurable benefits to patients with ESRD. The overall goal of this pilot trial is to evaluate the feasibility of conducting a randomized controlled trial of intensive vs liberalized phosphate control among hemodialysis recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 yrs
2. Receiving chronic hemodialysis for > 90 days,
3. Dialysis prescription is currently no more than 4 sessions per week and prescribed as 3-5 hrs per session
4. Most recent P value 1.30-2.50 mmol/L
5. Receipt of a calcium-based P binder

Exclusion Criteria:

1. Patient is booked (with a known surgical date) for a live donor kidney transplant in the next 26 weeks
2. Planned switch to a dialysis schedule that involves > 16 hours per week of therapy within the next 26 weeks.
3. Planned switch to peritoneal dialysis within the next 26 weeks
4. Pregnancy
5. Albumin-corrected serum calcium > 2.60 mmol/L in the past year requiring reduction of the calcium carbonate dose
6. History of calciphylaxis
7. Attending nephrologist believes that an otherwise eligible patient is mandated- on clinical grounds- to have a P value that is targeted to < 1.50 mmol/L or > 2.00 mmol/L
8. Attending nephrologist believes an otherwise eligible patient is not a candidate for escalation of the current calcium dose
9. Co-enrollment in a clinical trial where the intervention is deemed to interfere with the adherence, safety or efficacy of the intervention provided herein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Serum phosphate concentration | 26 weeks

SECONDARY OUTCOMES:
Number of patients who successfully achieved target serum P at week 26 based on the arm to which they were randomized | 26 weeks
Treatment compliance as defined by taking the study medication at least 80% of the time | 26 weeks
Number of serious adverse events | 26 weeks
Number of hospitalizations for vascular reasons that are unrelated to dialysis access | 26 weeks
Proportion of patients with a vascular death or non-fatal vascular event | 26 weeks
Proportion of patients developing serum calcium > 2.60 mmol/L | 26 weeks
Number of fractures | 26 weeks
Number of patients developing calcific uremic arteriolopathy (ie, calciphylaxis) | 26 weeks
Change in quality-of-life | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wald, MDCM, Principal Investigator — Unity Health Toronto
Locations (5):
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Capital District Health Authority, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario